CLINICAL TRIAL: NCT01970839
Title: Effect of Tourniquet on Sensory Nerve Conduction Threshold (sNCT) and OxyNeuroGram (ONG) Index- A Volunteer Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00048542
Record Dates: First submitted 2013-10-17; First posted 2013-10-28 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2016-08

CONDITIONS: Sensory Nerve Conduction; Oxyneurogram Index
Keywords: Tourniquet; Endoneural; Ischemia
MeSH Terms: conditions — Ischemia | interventions — Tourniquets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tourniquet, pain, nerve injury, sensory nerve function (Other)
  Interventions: Device: tourniquet, sensory nerve conduction abnormality

INTERVENTIONS:
Device: tourniquet, sensory nerve conduction abnormality

SUMMARY:
There are a number of risk factors for development of chronic pain that have been evaluated including age, gender, type and duration of surgery, duration of pain prior to surgery and tourniquet application. There is some scientific evidence from animal studies demonstrating that prolonged tourniquet application can result in lack of oxygen supply to nerves, and subsequent nerve damage resulting in chronic pain. This theory has not been proven in humans. In this study the investigators will indirectly assess the evidence for abnormalities caused by tourniquet application on subjects' nerves using well established devices to determine the function of these nerves.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Over 18 years of age

Exclusion Criteria:

* Neurological disease
* Diabetes mellitus
* History of nerve injury
* Chronic pain
* Alcoholism
* Blood pressure measurements greater than 140/80 and infection in the monitored area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Changes in sensory nerve conduction | baseline, 5 minutes
Changes in oxyneurogram index | baseline, 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Srini Pyati, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided